CLINICAL TRIAL: NCT03976570
Title: The Effect of Occupational Therapy on Subthreshold Attention Deficit Hyperactivity Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erzurum Regional Training & Research Hospital (Other Government)
Responsible Party: Principal Investigator, Hicran Doğru, Dr., Erzurum Regional Training & Research Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0001
Record Dates: First submitted 2019-06-04; First posted 2019-06-06 (Actual); Last update posted 2019-06-06 (Actual); Status verified 2019-06

CONDITIONS: Attention Deficit and Disruptive Behavior Disorders
MeSH Terms: conditions — Attention Deficit and Disruptive Behavior Disorders | interventions — Occupational Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Occupational Therapy (Experimental): Occupational Therapy
  Interventions: Behavioral: Occupational Therapy

INTERVENTIONS:
Behavioral: Occupational Therapy — Occupational therapy to children with subthreshold attention deficit hyperactivity disorder

SUMMARY:
The purpose of this study is to investigate the effectiveness of occupational therapy in subthreshold attention deficit hyperactivity disorder.

DETAILED DESCRIPTION:
Subthreshold attention deficit hyperactivity disorder may occur in a subset of children who are possibly more sensitive to their environment. Therefore, it is very important to target the elimination of symptoms with appropriate preventive therapies before this disorder occurs. One of the promising preventive therapy option may be occupational therapy.

Attention deficit hyperactivity disorder can have a negative impact on occupational performance such as: activities of daily living, education, resting, sleeping, playing and social participation. Occupational therapists are able to provide interventions to improve engagement in daily activities on social skills, play, executive functioning, impulsivity, inattention, and motor coordination.

Although the guidelines about the treatment of ADHD are primarily medically and psychologically based, certain treatment components are useful for occupational therapy practice; for example, behavioural management of the child and psychoeducational programmes for families.

However, treatment recommendations for subthreshold ADHD cases or the population at risk are limited. This study investigates the effectiveness of occupational therapy in subthreshold attention deficit hyperactivity disorder.

ELIGIBILITY:
Inclusion Criteria:

* Subthreshold Attention Deficit Hyperactivity Disorder

Exclusion Criteria:

* Attention Deficit Hyperactivity Disorder

Ages: 7 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2018-01-17 (Actual); Primary Completion 2018-07-17 (Actual); Study Completion 2018-07-17 (Actual)

PRIMARY OUTCOMES:
Dunn Sensory Profile | 12 weeks
  The Sensory Profile is a 125-item questionnaire filled out by the caregiver that describe responses to sensory events in daily life. It is a 5-point Likert scale how frequently the child uses that response to particular sensory events. This instrument evaluates the possible effects of sensory processing to a child's performance.
K-SADS-PL | 12 weeks
  The K-SADS-PL is a semi-structured interview scale, which is widely used and enables evaluation in 20 different diagnostic domains.

SECONDARY OUTCOMES:
The Conner's parent rating scale | 12 weeks
  The Conner's parent rating scale-revised: short form (CPRS-R:S): This standard measure is used as a diagnostic tool of Attention Deficit Hyperactivity Disorder. It consists of 27 items, each rated on a 4-point Likert scale (0=not true at all to 3=very much true). It has four subscales which are oppositional, hyperactivity, cognitive problems and ADHD index.
Conners' Teacher Rating Scale | 12 weeks
  Conners' Teacher Rating Scale- revised: short form (CTRS-R:S): This is a commonly used measure of behavioral problems associated with ADHD, which originally was developed as a measure of behavioral change for pharmacological studies. It is also 28 items (sixteen overlap with the original short-form). The CTRS-R:S has three scales which are Oppositional, Cognitive Problems/Inattention, and Hyperactivity.
Canadian Occupational Performance Measure | 12 weeks
  The Canadian Occupational Performance measure (COPM) is an outcome measure and semi-structured interview. It is a measure for identify goals in the areas of self-care, productivity and leisure/play that they have difficulty performing. In this study, each child selected three to five goals, and then parents and children rated performance and satisfaction on all goals using a 10-point scale. Changes in scores on baseline and end of therapy are determined separately. An increase of two or more points indicates clinically significant change.
Clinical Global Impressions (CGI) Scale: | 12 weeks
  The CGI scale was developed for use in clinical trials to provide a brief assessment of the clinician's view of the patient's functioning. The CGI has two components-the CGI-Severity (CGI-S), which rates illness severity (1=normal, not at all ill; 2=borderline mentally ill; 3=mildly ill; 4=moderately ill; 5=markedly ill; 6=severely ill; 7=among the most extremely ill) and the CGI-Improvement(CGI-I) (1=very much improved; 2=much improved; 3=minimally improved; 4=no change from baseline; 5=minimally worse; 6= much worse; 7=very much worse) which rates change from the initiation of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Hicran Doğru, Principal Investigator — Erzurum Regional and Training Hospital
Locations (1):
- Erzurum Regional Training and Research Hospital, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No